CLINICAL TRIAL: NCT05489848
Title: Chemotherapy Versus Chemoradiotherapy on the Prognosis for Postoperative Endometrial Cancer With P53-mutation Profile: a Non-inferiority Randomized Controlled Trial
Brief Title: Chemotherapy vs Chemoradiotherapy for Post-operative Endometrial Cancer Patients With P53-mutation
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yulan Ren, M.D, Ph.D, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC-2022 -01
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Paclitaxel; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1: Chemotherapy group (Experimental): Paclitaxel plus carboplatin (TC) regimen, intravenous chemotherapy. Once every three weeks with total of 6 cycles.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- Arm2: Radiotherapy plus chemotherapy group (Active Comparator): Stage IA: TC(Paclitaxel plus carboplatin) regimen for 4 course+/-VBT.
  Stage IB-II ( with no residual disease): TC regimen for 2 course +EBRT (external irradiation radiotherapy) plus cisplatin concurrent chemotherapy +TC regimen for 2 course ±VBT.
  Stage III-IVA ( with no residual disease) and any stage except IVB (residual disease <2cm): TC regimen for 2 course +EBRT (external irradiation radiotherapy) plus cisplatin concurrent chemotherapy +TC regimen for 2 course ±VBT.
  Radiotherapy can be started 3 weeks after the completion of the chemotherapy, and Chemotherapy can be started 2 - 3 weeks after the completion of radiotherapy.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Radiation: EBRT; Radiation: VBT

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel: paclitaxel dose of 135~175mg / m2, about 3 hours after the infusion, the use of pretreatment drugs before the infusion according to the drug instructions. Every 21 days is one session.
Drug: Carboplatin — Carboplatin: Doses were given at AUC=5 - 6 and used after paclitaxel. Based on the calculated amount, the maximum dose of carboplatin per chemotherapy does not exceed 750mg.
Drug: Cisplatin — Concurrent cisplatin intravenous chemotherapy on radiotherapy days 1 and 29,50mg / m2, a total of 2 times.
  Arms: Arm2: Radiotherapy plus chemotherapy group
Radiation: EBRT — 50.4Gy/28 / 6 weeks; common iliac node positive or paraaortic node positive plus extended field.The radiation extension field should include the entire pelvic cavity, the common iliac vessels and the paraaortic lymph node area.The range above the extension field is determined based on the clinical status, but at least 1-2cm above the renal vascular level.
  Arms: Arm2: Radiotherapy plus chemotherapy group
Radiation: VBT — Subnormal vaginal mucosa was 0.5cm, 30Gy / 5times /5weeks.
  Arms: Arm2: Radiotherapy plus chemotherapy group

SUMMARY:
Aim to compare chemotherapy alone or chemoradiotherapy for post-operative endometrial cancer (stage I-IVA) with p53 mutation.

DETAILED DESCRIPTION:
According to tumor molecular characteristic, endometrial cancer can be divided into four types with different biological behaviors and prognosis: POLE hypermutation （POLEmut）, Mismatch repair system defect (MMRd), Non special molecular feature (NSMP) and P53 mutation (p53mut) For the postoperative therapy, preliminary data showed that p53mut endometrial cancer was more sensitive to chemotherapy. Therefore, we propose a hypothesis: for p53mut endometrial carcinoma, compared with chemoradiotherapy, postoperative chemotherapy alone had similar effects on the prognosis and similar treatment-related adverse reactions, but could avoid radiotherapy-related adverse effects and reduce medical expenses. And more high-quality evidence is needed to prove the hypothesis.

This study were approved by the Fudan University Shanghai Cancer Center and all other institutes. Before initiation of study procedures, written informed consent will be obtained from each patient regarding risks of treatments and agreement of using their clinical data for research purpose.

Patients will be stratified into 4 layers by surgical pathological staging (FIGO 2009), preoperative and postoperative imaging evaluation, surgical conditions and postoperative pathology : stage IA,stage IB-II, stage III-IVA ( no residual lesion after operation), any stage with maximum diameter of residual lesion <2cm (except stage IVB). After stratification, Eligible patients in each stratification of each center will be randomly assigned (1:1) to receive:

Arm1:Paclitaxel plus carboplatin (TC) regimen, intravenous chemotherapy. Once every three weeks, a total of 6 course.

Arm2: Stage IA: TC regimen for 4 course+VBT. Stage IB-IVA (no residual lesion after operation) and any stage with maximum diameter of residual lesion <2cm (except stage IVB): TC regimen for 2 course +EBRT (external irradiation radiotherapy) plus cisplatin concurrent chemotherapy +TC regimen for 2 course (same as above) ±VBT.

The specific implementation plan should be performed after NCCN(2022 V1.) and ESGO guidelines, and adjuvant therapy is preferably started within 4-6 weeks after surgery and no later than 8 weeks after surgery.

The main research indicators of this study: PFS at 2 years after operation. Secondary research indicators: 3 years postoperative PFS and 5 years postoperative PFS and OS; adverse effects; quality of life; medical expenses; site of recurrence. And expression of molecular markers: Explore the correlation between the expression of molecular markers involved in IHC proteomics and molecular typing gene mutation detection of tumor tissue and therapeutic efficacy.

This study is an open label randomized controlled trial with non-inferiority design.Statistical analyses On the basis of data from previous studies (PORTEC-3, GOG-258, GOG-249 and Molecular Classification Of G3 EEC, etc.), the 2-year PFS of radiochemotherapy group is expected to be 75%, if that in chemotherapy-alone group was 65% and above,this group should not to be considered to be inferior, and the unilateral α level is 0.05, 80% of the detection efficiency. After patient stratification in each center, two groups were allocated by 1:1, with 15% total withdrawal groups and lost follow up rates, with an expected recruitment for 5 years and 5 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1)Age ≥18 years,

  2) Patients with stage I-IVA (FIGO2009) (excluded endometrial epithelial carcinoma confined to the endometrial layer), which have received initial diagnosis and comprehensive staging surgery (based on total uterine and double salpingectomy. Lymph nodes are evaluated by at least a sentinel lymph node biopsy), regardless of the pathological type, at the same time, the molecular typing of preoperative endometrial biopsy or total hysterectomy should be type p53mut.

  3)The duration of postoperative adjuvant therapy after initiation shall not exceed 8 weeks after enrollment,

  4)There is no obvious abnormality in the function of important organs, and the relevant test values meet the following requirements:

A. White blood cell count ≥3×109/L or absolute value of neutrophile granulocyte ≥ 1.5×109/L,

B. Platelet count ≥ 100× 109/L,

C. AST and/or ALT<2.5 times the upper limit of normal value,

D. Serum creatinine < 2 times the upper limit of normal value,

E. Physical fitness score: Karnofsky(KPS) score ≥60, The Eastern Cooperative Oncology Group(ECOG) score is ≤2 points.

Exclusion Criteria:

* 1) Tumors from uterine stroma,

  2) Recurrent endometrial malignant tumor,

  3) Those who have received other anti-tumor treatments within half a year before surgery: including neoadjuvant chemotherapy, hormone therapy, target therapy, immunotherapy, and biological therapy,etc.

  4) Those in pregnancy and perinatal period,

  5) Concurrent with other malignant tumors of reproductive system or non-reproductive system,

  6) History of important organ transplantation,

  7) Those who need to take immunosuppressants with a history of immune diseases,

  8) History of severe mental illness and brain dysfunction,

  9) History of drug abuse or drug use,

  10) Participants in other clinical trials at the same time,

  11) Those who are unable or unwilling to receive postoperative adjuvant chemotherapy or radio-chemotherapy/sign the informed consent form/comply with the research requirements,

  12) Patients of any stage who are excluded or unable to tolerate radiotherapy and chemotherapy after evaluation without indication of radiotherapy.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2022-08-20 (Estimated); Primary Completion 2028-08-20 (Estimated); Study Completion 2030-08-20 (Estimated)

PRIMARY OUTCOMES:
the 2-year progression-free survival(PFS) | 2 years
  The percentage of patients who have first relapse within 2 years after surgery.

SECONDARY OUTCOMES:
the 3-year PFS | 3 years
  The percentage of patients who have first relapse within 3 years after surgery.
the 5-year PFS and Overall survival(OS) | 5 years
  The percentage of patients who have first relapse within 5 years after surgery. The percentage of patients who died within 5 years after surgery.

OTHER OUTCOMES:
Incidence of adverse events | From date of recruitment, assessed up to 1 month after treatment.
  Adverse events related with intervention. Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v5.0 will be recorded, as well as incidence of adverse events.
Quality of life change | baseline, 6 months, 12 months
  Collect the questionnaire ETRTC-QLQ-C30 V3.0-EN, and count scores change through intervention (Chemotherapy or Radiochemotherapy)
Medical expenses | 5 years
  Medical expenses refer to all kinds of expenses incurred by patients in order to treat diseases. It includes not only the medical expenses and surgical expenses of doctors, but also the expenses of hospitalization, nursing, hospital equipment, etc.
Site of recurrence | 5 years
  The frequency of recurrence site in different groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yulan Ren, Principal Investigator — Fudan University; Huaying Wang, Principal Investigator — Fudan University